CLINICAL TRIAL: NCT01431534
Title: A Phase I Study of Ridaforolimus in Pediatric Patients With Advanced Solid Tumors
Brief Title: A Study of Ridaforolimus in Pediatric Participants With Advanced Solid Tumors (MK-8669-056)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8669-056; 2011-000729-55 (EudraCT Number); MK-8669-056 (Other: Merck Protocol Number)
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Solid Tumors
MeSH Terms: interventions — ridaforolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ridaforolimus 22 mg/m^2 (Experimental): Participants receive 22 mg/m^2 of ridaforolimus administered orally for 5 consecutive days each week (2 days rest) in consecutive 28-day cycles for up to six months. Eligible participants can receive additional treatment in an extension phase of the study.
  Interventions: Drug: Ridaforolimus
- Ridaforolimus 28 mg/m^2 (Experimental): Participants receive 28 mg/m^2 of ridaforolimus administered orally for 5 consecutive days each week (2 days rest) in consecutive 28-day cycles for up to six months. Eligible participants can receive additional treatment in an extension phase of the study.
  Interventions: Drug: Ridaforolimus
- Ridaforolimus 33 mg/m^2 (Experimental): Participants receive 33 mg/m^2 of ridaforolimus administered orally for 5 consecutive days each week (2 days rest) in consecutive 28-day cycles for up to six months. Eligible participants can receive additional treatment in an extension phase of the study.
  Interventions: Drug: Ridaforolimus

INTERVENTIONS:
Drug: Ridaforolimus — Oral administration of 10 mg enteric-coated tablets at doses of 22 mg/m^2, 28 mg/m^2, or 33 mg/m^2 based on body surface area (BSA), once daily for 5 consecutive days each week in consecutive 28-day cycles.
  Other Names: MK-8669

SUMMARY:
The main objectives of this trial are to determine the recommended dose of ridaforolimus for pediatric participants with advanced solid tumors by measuring the number of participants experiencing dose-limiting toxicities (DLTs) while on different doses of ridaforolimus, and to characterize the pharmacokinetics of ridaforolimus in these participants. The primary hypotheses of this study are that 1) the DLTs observed will be dose-dependent and allow for definition of a maximum tolerated dose (MTD) and 2) at a safe and well tolerated dose, ridaforolimus geometric mean (GM) Day-5 blood area under the concentration-time curve at 24 hours (AUC0-24) exceeds 75% (or 1304-ng*hr/mL) of the estimated GM Day-5, 40-mg AUC0-24 in adults.

Study-related visits concluded in August 2013. Participants who did not have disease progression, adequately tolerated therapy, and continued to meet eligibility criteria for 6 months after the enrollment period had been completed could continue treatment in an extension phase until they met discontinuation criteria or voluntarily withdrew.

ELIGIBILITY:
Inclusion criteria:

* Histologic or cytologic diagnosis of a malignant solid tumor, including tumors of the central nervous system and lymphoma, that have progressed despite standard therapy or for which no effective standard therapy is known. Participants who have received standard therapy and continue to have biopsy-proven residual stable disease are eligible
* Measurable or non-measurable disease
* Must be able to swallow tablets
* Performance Status: Lansky Play Scale ≥70 for children <10 years of age; Karnofsky score ≥70 for children ≥10 to <16 years; or Eastern Cooperative Oncology Group (ECOG) Status 0-2 for patients age 16 and older
* Adequate organ function
* For females of reproductive potential, a negative pregnancy test must be documented within 72 hours of receiving the first dose of study medication
* Participants of reproductive potential must agree to use (or have their partner use) adequate contraception throughout the study, starting with Visit 1 through 30 days after the last dose of study drug

Exclusion criteria:

* Currently receiving any other investigational agents or using any investigational devices
* Leukemia
* Participant previously received ridaforolimus, rapamycin, or other rapamycin analogs
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ridaforolimus
* Persistent acute toxicity from previous therapy ≥Grade 2 (excluding alopecia, neuropathy, or hearing loss)
* Uncontrolled intercurrent illness despite adequate therapy
* Pregnant or breastfeeding
* Requirement for concurrent treatment with medications that are inducers or inhibitors of cytochrome P450 (CYP3A)
* Poorly controlled Type 1 or 2 diabetes

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-01-30 (Actual); Primary Completion 2013-08-20 (Actual); Study Completion 2018-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Pearson AD, Federico SM, Aerts I, Hargrave DR, DuBois SG, Iannone R, Geschwindt RD, Wang R, Haluska FG, Trippett TM, Geoerger B. A phase 1 study of oral ridaforolimus in pediatric patients with advanced solid tumors. Oncotarget. 2016 Dec 20;7(51):84736-84747. doi: 10.18632/oncotarget.12450. PMID 27713169

RESULTS

PARTICIPANT FLOW:
Groups:
- Ridaforolimus 22 mg/m^2: Participants received 22 mg/m^2 of ridaforolimus administered orally for 5 consecutive days each week (2 days rest) in consecutive 28-day cycles for up to six months. Eligible participants could receive additional treatment in an extension phase of the study.
- Ridaforolimus 28 mg/m^2: Participants received 28 mg/m^2 of ridaforolimus administered orally for 5 consecutive days each week (2 days rest) in consecutive 28-day cycles for up to six months. Eligible participants could receive additional treatment in an extension phase of the study.
- Ridaforolimus 33 mg/m^2: Participants received 33 mg/m^2 of ridaforolimus administered orally for 5 consecutive days each week (2 days rest) in consecutive 28-day cycles for up to six months. Eligible participants could receive additional treatment in an extension phase of the study.
Period: Treatment Phase
Arm/Group | Ridaforolimus 22 mg/m^2 | Ridaforolimus 28 mg/m^2 | Ridaforolimus 33 mg/m^2
Started | 4 | 3 | 13
Completed | 0 | 0 | 2 (Participants completing Treatment Phase could continue in Extension Phase.)
Not Completed | 4 | 3 | 11
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Progressive Disease | 4 | 3 | 10
Period: Extension Phase
Arm/Group | Ridaforolimus 22 mg/m^2 | Ridaforolimus 28 mg/m^2 | Ridaforolimus 33 mg/m^2
Started | 0 (No participants continued in Extension Phase.) | 0 (No participants continued in Extension Phase.) | 2 (Participants from Treatment Phase who continued in Extension Phase.)
Completed | 0 | 0 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ridaforolimus 22 mg/m^2 | Ridaforolimus 28 mg/m^2 | Ridaforolimus 33 mg/m^2 | Total
Number analyzed (Participants) | 4 | 3 | 13 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.0 (5.7) | 14.7 (2.5) | 12.2 (3.3) | 12.8 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 8 | 12
  Male | 1 | 2 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Dose Limiting Toxicity (DLT) According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI-CTCAE v.4.0)
Description: DLT defined using NCI-CTCAE v.4.0 as any of the following events occurring during the first 28-day cycle that were possibly, probably, or definitely study drug-related: Grade 4 neutropenia for ≥5 days; Grade 3-4 neutropenia associated with fever, antibiotics, or hospitalization for infection; Grade 4 thrombocytopenia for ≥5 days or requiring platelet transfusion; ≥Grade 3 hyperglycemia for ≥5 days despite management; ≥Grade 3 diarrhea for >24 hours despite management; ≥Grade 3 nausea or vomiting despite management; any other Grade ≥3 non-hematological toxicity persisting despite management (except alopecia, transient electrolyte abnormalities, transient Grade 3 liver function test elevations, and Grade 3 neurotoxicity for participants with baseline Grade 3 neurotoxicity); inability to complete DLT assessment period, interruption in dosing for >10 dosing days during DLT assessment period, or any delay in the initiation of the next cycle for >10 dosing days due to any related toxicity.
Time Frame: Cycle 1 (cycle = 28 days)
Population: Participants who completed the first 28-day cycle of therapy with adequate drug exposure (>75% of planned study drug doses, exclusive of doses missed due to related toxicity), or who discontinued from the study due to a related DLT, were evaluable for DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Ridaforolimus 22 mg/m^2 | Ridaforolimus 28 mg/m^2 | Ridaforolimus 33 mg/m^2
Number analyzed (Participants) | 4 | 3 | 13
Participants | 0 | 0 | 1

2. Primary Outcome: Area Under the Concentration-Time Curve of Ridaforolimus From Time 0 to 24 Hours (AUC0-24 hr)
Description: AUC is a measure of the amount of drug in the blood over time. Whole blood samples were collected pre-dose (within 5 minutes of ridaforolimus administration) and post-dose at specified time points on Day 5 of the first week of Cycle 1 to determine AUC0-24 hr.
Time Frame: Day 5 of Cycle 1 [28-day cycle]: pre-dose (0.0 hours) and 0.5, 1.0, 2.0, 4.0, 8.0, and 24.0 hours after administration of ridaforolimus
Population: Participants who received all 5 ridaforolimus doses in the first week of 28-day Cycle 1 were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Ridaforolimus 22 mg/m^2 | Ridaforolimus 28 mg/m^2 | Ridaforolimus 33 mg/m^2
Number analyzed (Participants) | 4 | 3 | 11
hr*ng/mL | 1340 (31.7) | 2330 (36.2) | 2280 (29.8)

ADVERSE EVENTS:
Time Frame: Up to the 17-Dec-2013 database lock (up to ~56 weeks)
Description: All participants who received at least one dose of study treatment on the base study. Per protocol, safety data from the extension period were not included in the study database and did not contribute to the primary safety analysis.
Arm/Group | Ridaforolimus 22 mg/m^2 | Ridaforolimus 28 mg/m^2 | Ridaforolimus 33 mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/3 | 1/13
Serious Adverse Events (participants affected / at risk) | 3/4 | 2/3 | 7/13
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ridaforolimus 22 mg/m^2 (N=4) | Ridaforolimus 28 mg/m^2 (N=3) | Ridaforolimus 33 mg/m^2 (N=13)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ridaforolimus 22 mg/m^2 (N=4) | Ridaforolimus 28 mg/m^2 (N=3) | Ridaforolimus 33 mg/m^2 (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 3 (6)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 1 (1) | 3 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Mydriasis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 1 (1) | 2 (2)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 6 (11)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6) | 2 (2) | 8 (11)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 3 (4) | 10 (18)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (12) | 1 (1) | 7 (10)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 3 (3) | 7 (8)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 1 (2) | 4 (4)
Thrombosis in device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (4) | 1 (1) | 9 (15)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 2 (2) | 8 (15)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 4 (5)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 3 (4)
Blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 5 (8)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 6 (6)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood magnesium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 4 (8)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 1 (6) | 1 (1) | 1 (3)
Blood selenium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (2) | 1 (2) | 4 (5)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 2 (2) | 5 (6)
Haemoglobin decreased (Investigations) | 1 (4) | 1 (2) | 2 (6)
International normalised ratio decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (5) | 0 (0) | 4 (5)
Neutrophil count decreased (Investigations) | 1 (4) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 1 (3) | 0 (0) | 10 (17)
Reticulocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 4 (4)
White blood cell count decreased (Investigations) | 1 (5) | 2 (3) | 4 (9)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (7)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 3 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3) | 1 (2) | 1 (6)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 4 (6)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (6) | 1 (2) | 6 (11)
Hyporeflexia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Enuresis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 6 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin striae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.